CLINICAL TRIAL: NCT04966884
Title: The Efficacy and Safety of JAK Inhibitor in the Treatment of Anti-MDA5 Antibody-positive Dermatomyositis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-193
Record Dates: First submitted 2021-07-15; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Dermatomyositis, Adult Type
Keywords: Dermatomyositis,Tofacitinib,anti-MDA5 antibody
MeSH Terms: conditions — Dermatomyositis | interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-arm open-label pilot observational study (Experimental): Patients were received a glucocorticoids (0.8mg-1mg/kg/day) and a combination with tofacitinib (at a dose of 5 mg twice daily).
  Interventions: Drug: JAK Inhibitor

INTERVENTIONS:
Drug: JAK Inhibitor — 1. Prednisone 0.8-1.0 mg/kg/d, the dose was gradually reduced, and after 4 weeks, the dose was reduced by 5mg every two weeks, and then reduced to 10mg/d for 4-6 months after oral administration for 3 months, and then reduced to 7.5mg/d for maintenance therapy until 12 months;
  2. Tofacitinib 5 mg twice daily for 12 months.

SUMMARY:
Anti-melanoma differentiation-associated gene5 (Anti-MDA5) antibody positive Dermatomyositis (DM) is a subtype of DM that is more frequent in East Asia, which is often exhibit skin lesion, clinically amyopathic and interstitial lung disease. About 42%-100% of patients with Anti-MDA5+ DM develop rapidly progressive interstitial lung disease (RPILD) and result in respiratory failure. The mortality is as high as 40% within 6 months. In addition, not every patient with Anti-MDA5+ DM respond to traditional treatment strategy and most of the patients are resistant to immunosuppressive therapy including a combination of high dose glucocorticoids (GCs) and immunosuppressants such as cyclosporine, tacrolimus, or cyclophosphamide. However, RP-ILD is still the main cause of death due to fatal respiratory failure. Therefore, treatment of Anti-MDA5+ DM patients is challenging.Blocking multiple cytokines may become a new target for the treatment of this disease.Jakinibs is a Janus kinase (JAK) inhibitor that blocks a variety of cytokines, such as type I and type II interferon. Few studies have reported a positive response to JAK inhibitor for Anti-MDA5+ DM. Kazuhiro et al. reported in 2018 that JAK inhibitor tofacitinib may be an effective treatment option for high risk amyopathic dermatomyositis (ADM) -ILD patients after failure of conventional treatment, but the number of cases is too small. And a recent paper showed that great efficacy of tofacitinib for the improvement of survival of anti-MDA5-positive early-stage ADM-ILD patients.The aim of this study is to evaluate the efficacy and safety of JAK inhibitors in the treatment of anti-MDA5+ DM patients, and to evaluate the effect of JAK inhibitors on B cells of these patients, so as to provide a new target and theoretical basis for the treatment of anti-MDA5+ DM.

DETAILED DESCRIPTION:
Dermatomyositis (DM) is an idiopathic inflammatory myopathy characterized by chronic inflammation in the skin and muscle. Anti-melanoma differentiation-associated gene5 (Anti-MDA5) antibody positive DM is a subtype of DM that is more frequent in East Asia, which is often exhibit skin lesion, clinically amyopathic and interstitial lung disease. About 42%-100% of patients with Anti-MDA5+ DM develop rapidly progressive interstitial lung disease (RPILD) and result in respiratory failure. The mortality is as high as 40% within 6 months. In addition, not every patient with Anti-MDA5+ DM respond to traditional treatment strategy and most of the patients are resistant to immunosuppressive therapy including a combination of high dose glucocorticoids(GCs) and immunosuppressants such as cyclosporine, tacrolimus, or cyclophosphamide. However, RP-ILD is still the main cause of death due to fatal respiratory failure. Therefore, treatment of Anti-MDA5+ DM patients is challenging.The excessive production of multiple cytokines plays a crucial role in the development of Anti-MDA5+ DM patients complicated with ILD. Hyperferritinemia is a predictor of poor prognosis. Other abnormalities included lymphopenia, increased erythrocyte sedimentation rate(ESR), and elevated serum interleukin-18 (IL-18).Moreover, compared with Anti-MDA5- DM patients, serum interferon--α(IFN-α) concentration increased in Anti-MDA5+ DM patients with RP-ILD. Therefore, blocking multiple cytokines may become a new target for the treatment of this disease.Jakinibs is a Janus kinase (JAK) inhibitor that blocks a variety of cytokines, such as type I and type II IFN. Few studies have reported a positive response to JAK inhibitor for Anti-MDA5+ DM. Kazuhiro et al. reported in 2018 that JAK inhibitor tofacitinib may be an effective treatment option for high risk amyopathic dermatomyositis (ADM) -ILD patients after failure of conventional treatment, but the number of cases is too small. And a recent paper showed that great efficacy of tofacitinib for the improvement of survival of anti-MDA5-positive early-stage ADM-ILD patients.The aim of this study is to evaluate the efficacy and safety of JAK inhibitors in the treatment of anti-MDA5+ DM patients, and to evaluate the effect of JAK inhibitors on B cells of these patients, so as to provide a new target and theoretical basis for the treatment of anti-MDA5+ DM.This was a single-arm open-label pilot observational study. Patients were received a glucocorticoids (0.8mg-1mg/kg/day) and a combination with tofacitinib (at a dose of 5 mg twice daily). Inactive disease was defined as meeting the following three criteria: CK≤200U/L, physician visual analogue scale(VAS) =0, and myositis disease activity assessment visual analog scales (MYOACT) scores =0. Otherwise, the disease condition was considered to be active.The primary endpoint was the number of responders by total improvement score (TIS) ,which defined according to 2016 American College of Rheumatology(ACR)-European League Against Rheumatism(EULAR) Criteria for clinical response for adult DM/polymyositis(PM), after treatment with tofacitinib for 12 months. A TIS (0-100), determined by summing scores in each International Myositis Assessment and Clinical Studies Group (IMACS) core set measures (CSM). Thresholds for minimal, moderate, and major improvement were ≥20, ≥40, and ≥60 points in the TIS. Secondary endpoints included safety measures and change from baseline in the following index: percentage of predicted FVC (FVC % predicted) and percentage of predicted DLCO (DLCO% predicted), the ferritin level, peripheral lymphocyte subsets.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilled the Bohan and Peter criteria;
* anti-MDA5 antibody positive;
* patients who were not receiving treatment, or previously diagnosed with anti- MDA5-positive DM, who did not use biological agents (including but not limited to rituximab, infliximab, adalimumab, etanercept, tofacitinib, etc.) at the time of screening, or who had stopped taking drugs for ≥3 months;

Exclusion Criteria:

* patients if they had other connective tissue diseases, an underlying cancer, a concomitant infection, or a liver aminotransferase level greater than 2 times the upper limit of the normal range.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
TIS | 12 months
  the number of responders by total improvement score

SECONDARY OUTCOMES:
FVC % predicted | 12 months
  percentage of predicted FVC
DLCO % predicted | 12 months
  percentage of predicted DLCO
Lung high resolution CT score | 12 months
  Lung high resolution CT score
Overall survival rate | 12 months
  Overall survival rate%
Infection rate | 12 months
  Infection rate%

CONTACTS AND LOCATIONS:
Overall Officials: Lan He, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Department of Rheumatology, the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kurtzman DJB, Vleugels RA. Anti-melanoma differentiation-associated gene 5 (MDA5) dermatomyositis: A concise review with an emphasis on distinctive clinical features. J Am Acad Dermatol. 2018 Apr;78(4):776-785. doi: 10.1016/j.jaad.2017.12.010. Epub 2017 Dec 9. PMID 29229575
- [Result] Huang K, Vinik O, Shojania K, Yeung J, Shupak R, Nimmo M, Avina-Zubieta JA. Clinical spectrum and therapeutics in Canadian patients with anti-melanoma differentiation-associated gene 5 (MDA5)-positive dermatomyositis: a case-based review. Rheumatol Int. 2019 Nov;39(11):1971-1981. doi: 10.1007/s00296-019-04398-2. Epub 2019 Aug 2. PMID 31375890
- [Result] Kurasawa K, Arai S, Namiki Y, Tanaka A, Takamura Y, Owada T, Arima M, Maezawa R. Tofacitinib for refractory interstitial lung diseases in anti-melanoma differentiation-associated 5 gene antibody-positive dermatomyositis. Rheumatology (Oxford). 2018 Dec 1;57(12):2114-2119. doi: 10.1093/rheumatology/key188. PMID 30060040
- [Result] Chen Z, Wang X, Ye S. Tofacitinib in Amyopathic Dermatomyositis-Associated Interstitial Lung Disease. N Engl J Med. 2019 Jul 18;381(3):291-293. doi: 10.1056/NEJMc1900045. No abstract available. PMID 31314977